CLINICAL TRIAL: NCT04421872
Title: The Relationship Between the Disorder of Circadian Clock Gene and Early Cognitive Dysfunction After General Anesthesia
Brief Title: The Disorder of Circadian Clock Gene and Early Cognitive Dysfunction After General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, Principal investigator, Shengjing Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: general anesthesia and POCD
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Delirium; General Anesthesia; Exosomes; Clock Gene; Circadian Rhythm Disorders
Keywords: Postoperative Delirium; general anesthesia; Exosomes; clock gene; Circadian Rhythm Disorders
MeSH Terms: conditions — Emergence Delirium; Chronobiology Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia Group (Experimental)
  Interventions: Other: receiving general anesthesia
- Healthy control group (No Intervention)

INTERVENTIONS:
Other: receiving general anesthesia — patients receiving surgery under general anesthesia
  Arms: General anesthesia Group

SUMMARY:
Postoperative cognitive dysfunction (POCD) is a common postoperative complication in patients aged 65 and over, which refers to cognitive function changes such as memory decline and attention deficit after anesthesia and surgery. In severe cases, personality changes and social behavior decline may also occur, resulting in irreversible cognitive impairment.Previous studies have suggested that cognitive dysfunction after general anesthesia is linked to a genetic disorder of the body clock.Exosomes are cellular forms of cellular microvesicles containing complex RNA and proteins.Exosomes can mediate the expression of genes in the late transcriptional period of the clock system, and directly or indirectly participate in the negative regulation of rhythm expression of minute control genes, playing an important role in the intercellular circadian rhythm information output pathway.Rhythm disorders in the core biological clock system of urinary exosomes and the clock control genes related to kidney can early indicate circadian rhythm changes in the core biological clock system.The sorting and detection of urinary exosome clock information materials in patients has the advantages of easy access, continuous monitoring, early diagnosis and less damage, making urinary exosome a biomarker for the diagnosis and monitoring of circadian rhythm of a good kidney biological clock system.

ELIGIBILITY:
Inclusion Criteria:

* patients whose age ≥ 18 years old and <90 years of preoperative sleep disorder;
* Primary cancer patients who had not received any radiotherapy or chemotherapy before surgery;
* Surgeries expected to be performed under general anesthesia after ≧3 hours

Exclusion Criteria:

* a history of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis;
* inability to communicate due to coma, severe dementia, language impairment or serious illness;
* critically ill (preoperative ASA (American Society of Anesthesiologists)>III), Childe-Pugh C or severe renal insufficiency (preoperative dialysis);
* Neurosurgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive testing | one day before the surgery
  Neurocognitive testing was performed preoperatively and 6 weeks postoperatively, followed up 1 and 3 years postoperatively.
Neurocognitive testing | 6 weeks after surgery
  Neurocognitive testing was performed preoperatively and 6 weeks postoperatively, followed up 1 and 3 years postoperatively.
Neurocognitive testing | 1 year after surgery
  Neurocognitive testing was performed preoperatively and 6 weeks postoperatively, followed up 1 and 3 years postoperatively.
Neurocognitive testing | 3 years after surgery
  Neurocognitive testing was performed preoperatively and 6 weeks postoperatively, followed up 1 and 3 years postoperatively.
Core clock gene and kidney clock control gene detection | at the end of surgery
  The urine exosomes were extracted by overspeed centrifugation method. The mRNA ( messenger ribonucleic acid) expression results of the core heart clock gene and the renal bell control genes in the urinary exosomes were detected by timing and quantitative PCR(Polymerase Chain Reaction) and the rhythm was analyzed
Blood samples and Apolipoprotein E genotyping | at the end of surgery
  peripheral blood was collected from each patient for apolipoprotein E genotyping.

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Zhu, Principal Investigator — Shengjing Hospital
Locations (1):
- Junchao Zhu, Shenyang, China

IPD SHARING:
Plan to Share IPD: No